CLINICAL TRIAL: NCT07233954
Title: Use of i.v. Sodium Fluorescein as a Fluorescent Intra-operative Tracer in Patients With Suspected Malignant Neoplasms of the CNS
Brief Title: Intraoperative Use of I.V. Sodium Fluorescein in Suspected CNS Tumors
Acronym: FLUOCERTUM
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: FLUO.CER.TUM
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: CNS
Keywords: Neurosurgical Procedures; Malignant Neoplasms; Surgical Margins; Fluorescein
MeSH Terms: conditions — Neoplasms; Margins of Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The FLUO.CER.TUM study is a prospective observational clinical trial conducted at the IRCCS Foundation Neurological Institute "Carlo Besta" in Milan, Italy. It investigates the intraoperative use of intravenous sodium fluorescein as a fluorescent tracer to assist in the surgical resection of suspected malignant tumors of the central nervous system (CNS). These tumors typically present as contrast-enhancing masses on pre-operative MRI or CT scans.

Malignant brain tumors are notoriously difficult to fully resect due to challenges in distinguishing tumor margins from healthy tissue. Sodium fluorescein, a dye that accumulates in areas where the blood-brain barrier is disrupted, offers a promising solution by enhancing tumor visualization during surgery. When used with a dedicated surgical microscope equipped with a fluorescence filter, fluorescein can help surgeons identify and remove more tumor tissue, potentially improving patient outcomes.

The study aims to evaluate the effectiveness and safety of fluorescein-guided surgery in a real-world clinical setting. Approximately 800 patients of any age and gender, with suspected aggressive CNS lesions, will be enrolled. Each patient will receive 5 mg/kg of sodium fluorescein intravenously at the induction of anesthesia. Surgery will be performed using fluorescence-guided techniques, and patients will undergo pre- and post-operative imaging to assess the extent of resection. Clinical and neurological evaluations will also be conducted to monitor outcomes and any adverse effects.

The primary objective is to qualitatively assess the intraoperative fluorescence characteristics of CNS tumors. Secondary objectives include measuring the extent of tumor resection, evaluating post-operative neurological function, and documenting any side effects related to fluorescein administration.

The study adheres to ethical standards, including informed consent and approval by an ethics committee, and will be conducted in accordance with Good Clinical Practice guidelines and the Declaration of Helsinki. Data will be anonymized and securely stored, with results potentially published following appropriate review and approval.

DETAILED DESCRIPTION:
This clinical study investigates the intraoperative use of intravenous sodium fluorescein as a fluorescent tracer to assist in the surgical resection of aggressive tumors of the central nervous system (CNS). These tumors typically present as contrast-enhancing masses on pre-operative MRI or CT scans. The study is conducted at the IRCCS Foundation Neurological Institute "Carlo Besta" in Milan and follows a prospective observational design.

Malignant CNS tumors are often difficult to completely remove due to the challenge of distinguishing tumor margins from healthy brain tissue. This limitation affects prognosis, especially in high-grade gliomas. Sodium fluorescein, a dye historically used in ophthalmology, accumulates in areas where the blood-brain barrier is disrupted-such as in aggressive brain tumors-making it a potentially ideal agent for enhancing intraoperative visualization. When used with a surgical microscope equipped with a dedicated fluorescence filter, fluorescein allows surgeons to better identify tumor tissue during resection.

The study includes approximately 800 patients of any age and gender, all presenting with suspected aggressive CNS lesions based on contrast-enhanced imaging. Each patient receives 5 mg/kg of sodium fluorescein intravenously at the induction of anesthesia. Surgery is performed using fluorescence-guided techniques, and patients undergo pre- and post-operative imaging to assess the extent of resection. Clinical and neurological evaluations are conducted before and after surgery, with follow-up extending to the third post-operative day.

The primary objective is to qualitatively assess the intraoperative fluorescence characteristics of CNS tumors. Secondary objectives include evaluating the extent of tumor resection based on early post-operative imaging, monitoring neurological outcomes, and documenting any adverse reactions to fluorescein. Safety parameters such as blood pressure, heart rate, oxygen saturation, temperature, and renal function are monitored according to guidelines from the Italian Medicines Agency (AIFA).

Ethical approval is obtained from the appropriate Ethics Committee, and all patients provide informed consent prior to participation. The study complies with Good Clinical Practice (GCP) and the Declaration of Helsinki. Data are anonymized and stored securely, and results may be published following review and approval by the involved parties.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders, at any age.
2. Patients with suspected aggressive lesion of the CNS, as suggested by pre-operative MRI or CT with i.v. contrast agent administration.

Exclusion Criteria:

1. Impossibility to give consent due to cognitive deficits or language disorder.
2. Known allergy to contrast agents and/or history of previous anaphylactic shocks.
3. Known severe previous adverse reactions to Fluorescein
4. Acute myocardial infarction or stroke in the last 90 days.
5. Severe renal failure;
6. Severe hepatic failure;
7. Women in their first trimester of pregnancy or lactation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both genders, at any age.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Fluorescence Characteristics: Fluorescence Intensity of CNS Tumors | During surgical procedure
  Fluorescence intensity of aggressive CNS tumors during surgery using sodium fluorescein and a dedicated surgical microscope.
  Metric: Visual intensity of fluorescence in relation to tumor margins (measured on a standardized scale).
Intraoperative Fluorescence Characteristics: Fluorescence Distribution of CNS Tumors | During surgery
  Fluorescence distribution of aggressive CNS tumors during surgery using sodium fluorescein and a dedicated surgical microscope.
  Metric: Spatial distribution of fluorescence relative to tumor margins (e.g., focal vs. diffuse)
Intraoperative Fluorescence Characteristics: Fluorescence Clarity of CNS Tumors | During surgery
  Fluorescence clarity of aggressive CNS tumors during surgery using sodium fluorescein and a dedicated surgical microscope.
  Metric: Sharpness/definition of fluorescence edges in relation to tumor margins (scored visually)

SECONDARY OUTCOMES:
Extent of Tumor Resection | Within 72 hours post-surgery
  Quantitative evaluation of the percentage of tumor removed, based on early post-operative MRI or CT with contrast.
  Metric: Volume of residual tumor compared to pre-operative imaging.
Post-operative Neurological Function | Within 72 hours post-surgery
  Description: Assessment of neurological status following surgery, including motor, sensory, and cognitive functions.
  Metric: Standard neurological examination scores.
Adverse Reactions to Fluorescein | Up to 3 days post-surgery
  Monitoring and documentation of any side effects or adverse events related to the administration of sodium fluorescein.
  Metric: Incidence and severity of adverse events (e.g., allergic reactions, renal/hepatic changes)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan A Broggi, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts DW, Hartov A, Kennedy FE, Miga MI, Paulsen KD. Intraoperative brain shift and deformation: a quantitative analysis of cortical displacement in 28 cases. Neurosurgery. 1998 Oct;43(4):749-58; discussion 758-60. doi: 10.1097/00006123-199810000-00010. PMID 9766300
- [Background] Rasmussen IA Jr, Lindseth F, Rygh OM, Berntsen EM, Selbekk T, Xu J, Nagelhus Hernes TA, Harg E, Haberg A, Unsgaard G. Functional neuronavigation combined with intra-operative 3D ultrasound: initial experiences during surgical resections close to eloquent brain areas and future directions in automatic brain shift compensation of preoperative data. Acta Neurochir (Wien). 2007;149(4):365-78. doi: 10.1007/s00701-006-1110-0. Epub 2007 Feb 19. PMID 17308976
- [Background] Ramirez C, Bowman C, Maurage CA, Dubois F, Blond S, Porchet N, Escande F. Loss of 1p, 19q, and 10q heterozygosity prospectively predicts prognosis of oligodendroglial tumors--towards individualized tumor treatment? Neuro Oncol. 2010 May;12(5):490-9. doi: 10.1093/neuonc/nop071. Epub 2010 Feb 14. PMID 20156805
- [Background] Pedersen MW, Meltorn M, Damstrup L, Poulsen HS. The type III epidermal growth factor receptor mutation. Biological significance and potential target for anti-cancer therapy. Ann Oncol. 2001 Jun;12(6):745-60. doi: 10.1023/a:1011177318162. PMID 11484948
- [Background] Ohue S, Kumon Y, Nagato S, Kohno S, Harada H, Nakagawa K, Kikuchi K, Miki H, Ohnishi T. Evaluation of intraoperative brain shift using an ultrasound-linked navigation system for brain tumor surgery. Neurol Med Chir (Tokyo). 2010;50(4):291-300. doi: 10.2176/nmc.50.291. PMID 20448420
- [Background] Kwan AS, Barry C, McAllister IL, Constable I. Fluorescein angiography and adverse drug reactions revisited: the Lions Eye experience. Clin Exp Ophthalmol. 2006 Jan-Feb;34(1):33-8. doi: 10.1111/j.1442-9071.2006.01136.x. PMID 16451256
- [Background] Koc K, Anik I, Cabuk B, Ceylan S. Fluorescein sodium-guided surgery in glioblastoma multiforme: a prospective evaluation. Br J Neurosurg. 2008 Feb;22(1):99-103. doi: 10.1080/02688690701765524. PMID 18224529
- [Background] Heimberger AB, Crotty LE, Archer GE, Hess KR, Wikstrand CJ, Friedman AH, Friedman HS, Bigner DD, Sampson JH. Epidermal growth factor receptor VIII peptide vaccination is efficacious against established intracerebral tumors. Clin Cancer Res. 2003 Sep 15;9(11):4247-54. PMID 14519652
- [Background] Hegi ME, Diserens AC, Godard S, Dietrich PY, Regli L, Ostermann S, Otten P, Van Melle G, de Tribolet N, Stupp R. Clinical trial substantiates the predictive value of O-6-methylguanine-DNA methyltransferase promoter methylation in glioblastoma patients treated with temozolomide. Clin Cancer Res. 2004 Mar 15;10(6):1871-4. doi: 10.1158/1078-0432.ccr-03-0384. PMID 15041700
- [Background] Hall WA, Truwit CL. Intraoperative magnetic resonance imaging. Acta Neurochir Suppl. 2011;109:119-29. doi: 10.1007/978-3-211-99651-5_19. PMID 20960331
- [Background] Gulati S, Berntsen EM, Solheim O, Kvistad KA, Haberg A, Selbekk T, Torp SH, Unsgaard G. Surgical resection of high-grade gliomas in eloquent regions guided by blood oxygenation level dependent functional magnetic resonance imaging, diffusion tensor tractography, and intraoperative navigated 3D ultrasound. Minim Invasive Neurosurg. 2009 Feb;52(1):17-24. doi: 10.1055/s-0028-1104566. Epub 2009 Feb 26. PMID 19247900
- [Background] Esposito V, Paolini S, Morace R, Colonnese C, Venditti E, Calistri V, Cantore G. Intraoperative localization of subcortical brain lesions. Acta Neurochir (Wien). 2008 Jun;150(6):537-42; discussion 543. doi: 10.1007/s00701-008-1592-z. Epub 2008 May 6. PMID 18458808
- [Background] Eoli M, Silvani A, Pollo B, Bianchessi D, Menghi F, Valletta L, Broggi G, Boiardi A, Bruzzone MG, Finocchiaro G. Molecular markers of gliomas: a clinical approach. Neurol Res. 2006 Jul;28(5):538-41. doi: 10.1179/016164106X116827. PMID 16808886
- [Background] Cairncross JG, Ueki K, Zlatescu MC, Lisle DK, Finkelstein DM, Hammond RR, Silver JS, Stark PC, Macdonald DR, Ino Y, Ramsay DA, Louis DN. Specific genetic predictors of chemotherapeutic response and survival in patients with anaplastic oligodendrogliomas. J Natl Cancer Inst. 1998 Oct 7;90(19):1473-9. doi: 10.1093/jnci/90.19.1473. PMID 9776413
- [Background] Albert FK, Forsting M, Sartor K, Adams HP, Kunze S. Early postoperative magnetic resonance imaging after resection of malignant glioma: objective evaluation of residual tumor and its influence on regrowth and prognosis. Neurosurgery. 1994 Jan;34(1):45-60; discussion 60-1. doi: 10.1097/00006123-199401000-00008. PMID 8121569